CLINICAL TRIAL: NCT01820884
Title: The Safety of Ovarian Preservation in Stage IA Endometrial Carcinoma: A Multicenter, Prospective, Randomized Trial
Brief Title: The Safety of Ovarian Preservation in Stage IA Endometrial Carcinoma
Acronym: EC-02
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ding Ma (Other)
Collaborators: Shandong University (Other); Huazhong University of Science and Technology (Other); Zhejiang University (Other)
Responsible Party: Sponsor-Investigator, Ding Ma, Director of the department of Obstetrics and Gynecology, Tongji Hospital, Huazhong University of Science and Technology
Organization: Huazhong University of Science and Technology (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-GYN/EC-02
Record Dates: First submitted 2013-03-21; First posted 2013-03-29 (Estimated); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Endometrial Neoplasms
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Total Hysterectomy (TH) (Experimental): Patients may receive total hysterectomy (TH) and bilateral pelvic and para-aortic lymph node dissection (BPLND).
  Interventions: Procedure: TH; Procedure: BPLND
- TH and bilateral salpingo-oophorectomy (TH/BSO) (Active Comparator): Patients may receive total hysterectomy, bilateral salpingo-oophorectomy (BSO) and bilateral pelvic and para-aortic lymph node dissection.
  Interventions: Procedure: TH/BSO; Procedure: BPLND

INTERVENTIONS:
Procedure: TH — Total hysterectomy
  Arms: Total Hysterectomy (TH)
Procedure: TH/BSO — Total hysterectomy and bilateral salpingo-oophorectomy
  Arms: TH and bilateral salpingo-oophorectomy (TH/BSO)
Procedure: BPLND — bilateral pelvic and para-aortic lymph node dissection

SUMMARY:
This randomized trial is studying the efficacy and safety of the hysterectomy alone compared with hysterectomy and bilateral salpingo-oophorectomy (BSO) for patients with Stage IA endometrial carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* FIGO stage: ⅠA, endometrial carcinoma;
* Female, Chinese women;
* premenopausal women；
* ≤ 50 years old;
* Pathological diagnosis by curettage/hysteroscopy : G1
* No prior treatment;
* Provide written informed consent.

Exclusion Criteria:

* The suspicious metastasis of ovarian;
* Family history of ovarian cancer;
* Suffering from other malignancies;
* Concurrently participating in other clinical trials;
* Unable or unwilling to sign informed consents;
* Unable or unwilling to abide by protocol.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 240 (Estimated)
Dates: Start 2012-11; Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival (DFS) | 3-year DFS

SECONDARY OUTCOMES:
Clinical gynecologic endocrine function | 1-year period
  To observe the level of female hormone，i.e., estrogen, FSH, LH
Quality of Life | 3-year period
Overall Survival (OS) | 3-year OS

CONTACTS AND LOCATIONS:
Overall Officials: Beihua Kong, MD, PhD, Study Chair — Shandong University
Locations (3):
- China (3):
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Qilu Hospital，Shandong University, Jinan, Shandong
  - Women's Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang